CLINICAL TRIAL: NCT03488472
Title: A Pilot and Feasibility Trial to Determine the Rate of the Brain Relapse in Small Cell Lung Cancer (SCLC) Patients With Brain Metastases Treated With Stereotactic Radiosurgery (SRS) Followed by Tumor Treating Fields (TTF)
Brief Title: Radiosurgery Plus NovoTTF-200A for Metastatic Small Cell Lung Cancer to the Brain
Acronym: RAD 1704
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This feasibility study only accrued one patient since site activation. We believe that the primary reason for this is low patient motivation to go on study and wear the device. We attempted to broaden this study to partner sites without success.
Sponsor: Drexell Hunter Boggs (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Drexell Hunter Boggs, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001201
Record Dates: First submitted 2018-03-28; First posted 2018-04-05 (Actual); Results first posted 2023-01-04 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Brain Metastases; Small Cell Lung Cancer
MeSH Terms: conditions — Brain Neoplasms; Small Cell Lung Carcinoma | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- NovoTTF-200A device + Stereotactic Radiosurgery (SRS) (Experimental): Patients will undergo SRS treatment followed by continuous TTFields by wearing the NovoTTF-200A device over 18 hours QD. Treatment continues for up to 1 year or until progression.
  Interventions: Device: NovoTTF-200A; Radiation: Stereotactic Radiosurgery (SRS)

INTERVENTIONS:
Device: NovoTTF-200A — Begins within 7 days of SRS and continues until progression, death, or unacceptable toxicity.
Radiation: Stereotactic Radiosurgery (SRS) — SRS will begin within 21 days of study enrollment for 5-6 Gy per fraction for a total of 25 or 30 Gy.

SUMMARY:
This study is a prospective single arm trial designed to study the safety and effectiveness of a medical device, NovoTTF-200A, used with stereotactic radiosurgery (SRS) in subjects with brain metastases from small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
Tumor Treating Fields (TTFields) are low intensity alternating electric fields, which are tuned to interfere with the division process of cancer cells. TTFields are delivered to the region of cancer using an investigational device, called the NovoTTF-200A system. The device is portable, light weighted, battery operated device designed to deliver TTFields to brain metastases from small cell lung cancer (SCLC).

TTFields are a novel, non-invasive regional anti-mitotic treatment modality. Pre-clinical studies and clinical data in glioblastoma multiforme (GBM) have demonstrated a favorable safety profile and clinical superiority when treating the brain with TTFields. In addition, durable response have been demonstrated with 200kHz TTFields monotherapy for supratentorial tumors of the brain.

The development of brain metastases is devastating for SCLC patients and their families. Treatment options in this setting are limited to SRS or WBRT or a combination thereof. Few clinicians treat SCLC brain metastases with SRS alone because intracranial recurrence is high due to the fact that the entire brain is not treated. WBRT treats the entire brain and improves intracranial control, but at the risk of neurocognitive complications. Thus, new therapeutic options are needed, particularly ones that allow for greater intracranial control while minimizing the risk of neurocognitive adverse events. As such, TTFields following SRS may allow for sufficient regional treatment of the brain to eliminate any remaining tumor cells following radiosurgery as well as micro-metastases that remain untreated, and ultimately prolong intracranial control. Due to the favorable safety profile seen in phase III recurrent and newly diagnosed glioblastoma trials and in which the patients reported improved neurocognitive and emotional functioning, NovoTTF-200A is not expected to have neuro-toxic effects seen with WBRT.

Thus, the investigators hypothesize that the use of NovoTTF-200A applied to the brain following SRS for SCLC brain metastases will have cerebral control comparable to WBRT with less neurocognitive effects.

The patient will undergo stereotactic radiosurgery (SRS). Radiosurgery is a single treatment and will be done as an outpatient procedure.

Stereotactic Radiosurgery (SRS) will be followed by continuous TTFields treatment using the NovoTTF-200A. The patient will start using the NovoTTF-200A device within 7 days of SRS. The NovoTTF-200A treatment will be started by the device support specialist (DSS), trained by NovoCure, or by your study doctor. The patient will be educated and trained on how to properly use the device in the clinic or by a separately scheduled home visit. During this visit, the patient will be told how to operate the device, replace depleted batteries, recharge them, and connect to an external power supply. All patients will be required to shave their head, so the transducer arrays can be placed. Patients will wear 4 electronically insulated transducer arrays (sticky pads) on the top of the patient's head (based on the patient's tumor location) for the time the patient is using the device.

After this visit, the patient will continue treatment at home where participants can maintain regular daily routine. The patient must use the device for at least 18 hours a day per day on average. Breaks are allowed for personal needs (e.g. showering/bathing, array exchange). Patients will be instructed to replace the Transducer arrays 2-3 times a week with help of a caregiver. Patients will be instructed to use the device for a minimum of 4 weeks from the time of initiation. The NovoTTF-200A device will be inspected, either by the study doctor, research nurse, or by a Novocure representative, on a monthly basis to assess the patient's compliance with treatment. Each course of using the device will consist of continuous NovoTTF-200A use for one month. Multiple courses will be offered as long as the patient's tumor(s) in the brain have not come back. If the patient's tumor(s) do come back, the patient will need to terminate use of NovoTTF-200A. If tumors do not return in the patient's brain, the patient will be able to stay on NovoTTF-200A for up to 1 year.

Patients will be asked to visit the study doctor for follow-up care at several monthly intervals (1, 3, 6, 9, an 12 months after completion of stereotactic radiosurgery), or until the tumor(s) in the patient's brain return.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have history of histologically confirmed small cell lung cancer. Brain biopsy is not required unless diagnosis is judged to be in doubt by the treating physician.
* Brain metastases that have not received radiotherapy previously (metastases on post-contrast MRI obtained within six weeks of study entry) deemed to be amenable to SRS.

  * Longest diameter < 4 cm
* Prior prophylactic cranial irradiation (PCI) is allowed. The maximum allowed dose is 25Gy in 10 fractions.
* Prior systemic therapy is allowed after diagnosis of brain metastases provided that restaging MRI shows measurable intracranial disease.
* Karnofsky Performance Status (KPS) of greater than or equal to 70.
* Age greater than or equal to 18 years.
* Life expectancy greater than 3 months.
* Must receive optimal therapy for extracranial disease and may continue on systemic therapy during TTF administration.
* Ability to operate the NovoTTF-200A device independently or with caregiver aid.
* Previous clinical trial enrollment is allowed.
* Subjects given written informed consent.

Exclusion Criteria:

* History of prior brain metastases.
* Patients with significant edema leading to risk of brain herniation.
* History of prior whole brain radiotherapy (WBRT) other than prophylactic cranial radiation. Prophylactic cranial radiation with a maximum dose of 25 Gy delivered as 10 fractions is allowed. WBRT in excess of 25 Gy (anything over 25 Gy) is not allowed.
* Diffuse Leptomeningeal metastases with radiographic involvement in the brain and/or spinal cord. This does not include local leptomeningeal involvement which is defined as leptomeningeal enhancement within direct contact of targetable metastases.
* Implantable electronic device in the brain.
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea, or reduced level of consciousness).
* Known allergies to medical adhesives or hydrogel.
* Currently pregnant or breastfeeding.
* Concurrent brain-directed therapy.
* Insufficient recovery from all active toxicities of prior therapies.
* Women of childbearing potential who are not using an effective method of contraception are excluded.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Drexell H Boggs, MD, Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (1):
- University of Alabama at Birmingham (UAB), Hazelrig-Salter Radiation Oncology Center (HSROC), Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
Started | 1
Completed | 0
Not Completed | 1
Not completed — disease progression additional mets | 1

BASELINE CHARACTERISTICS:
Population: Terminated early.
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Distant Metastases
Description: Rate of distant CNS metastases/progression will be calculated as the total number of patients with such events divided by the total number of patients.
Time Frame: From date of first SRS treatment to time of the 6 month follow-up MRI
Population: The 1 patient enrolled started treatment but was discontinued due adrenal mets. Therefore, data not collected.
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: Overall survival will be measured as time from first SRS treatment to date of death, or censored as the last follow-up, whichever comes first. Overall survival rates will be analyzed using the Kaplan-Meier (KM) method.
Time Frame: From time of first SRS treatment to date of death, or censored as the last follow-up, whichever comes first, for up to 1 year.
Population: The 1 patient enrolled started treatment but was discontinued due adrenal mets. Therefore, data not collected.
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 0

3. Secondary Outcome: Local Recurrence
Description: Local recurrence will be defined as a measurable lesion deemed likely to be a brain metastases found within the treated area.
Time Frame: as for outcome 2
Population: The 1 patient enrolled started treatment but was discontinued due adrenal mets. Therefore, data not collected.
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 0

4. Secondary Outcome: Distant CNS Progression
Description: Distant CNS Progression is defined as development of new metastases outside the treated area.
Time Frame: as for outcome 2
Population: The 1 patient enrolled started treatment but was discontinued due adrenal mets. Therefore, data not collected.
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | NovoTTF-200A Device + Stereotactic Radiosurgery (SRS)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The 1 patient enrolled started treatment but was discontinued due adrenal mets. Therefore, data not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03488472/Prot_SAP_000.pdf